CLINICAL TRIAL: NCT02047123
Title: Nutritional Intervention With Yogurt and Flaxseed in Women With Profiles Lipidic to the Limit: A Randomized Controlled Trial
Brief Title: Nutritional Intervention With Yogurt and Flaxseed in Women With Profiles Lipi
Acronym: flaxseed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Elena García García, PID, Universidad Miguel Hernandez de Elche
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Elena García-García 2; Enrique Roche Collado (Other Grant/Funding Number: Instituto de Salud Carlos III-FEDER PS09/01093)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Overweight
Keywords: commercial flaxseed; cholesterol; lipidic profile; yoghurt; consumption
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raw Flaxseed (Experimental): For 30 days, participants in group 1 took with 15g flaxseed mixed with yoghurt and diet,(the 15g of raw flaxseed that was provided in addition to the linen package spoon so all would take far it) group 2 took yoghurt and diet, and group 3 only received the diet.The energy intake of the designed diet was similar into the three groups (ranging 1900-2000 Kcal per day).
  Interventions: Dietary Supplement: Raw Flaxseed

INTERVENTIONS:
Dietary Supplement: Raw Flaxseed — The participants were randomly single blind controlled trial distributed into three groups: (1, n =30), (2, n =32), (3, n =27). For 30 days, participants in group 1 took with 15g flaxseed mixed with yoghurt and diet,(the 15g of flaxseed that was provided in addition to the linen package spoon so all would take far it) group 2 took yoghurt and diet, and group 3 only received the diet.
  Other Names: Raw Flaxseed "Lino Dorado" 8426904171561

SUMMARY:
Flax (Linum usitatissimum L.) is an economically important oilseed. Lifestyle and diet are the first line interventions to reduce the short-term and long-term cardiovascular risk factors. Due to its high content of lignans, α-linolenic acid (LNA) and fiber, flaxseed has a beneficial effect on CVD risk factors, components to decrease the risk of cardiovascular disease. Objective: To determine the effect of the consumption of flax seed yogurt on the women lipid profile values to the limit, users of a pharmacy in Elche and in this way reduce the small dyslipidemia. The investigators performed an intervention including 133 women (age= 25-70 years). Participants were randomly and double-blind distributed into three groups: Group 1 (n= 30) consumed flaxseed (FS), yoghurt (Y) and diet (D), Group 2 (n= 32) volunteers consumed (Y) + (D) and Group 3 (n=27) consumed only diet. All groups followed a limit levels-cholesterol diet. Circulating total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides and were determined at the beginning and end of a 30-day test. As a result, group 1 presented significantly reduced total cholesterol levels. Correlation analysis indicated that the intake of (FS) could explain the flaxseed effect of the variation of the cholesterol and TG in this group. Altogether, this study concludes that consumption FS exert a positive impact in total cholesterol level and TG

DETAILED DESCRIPTION:
It is an analytical intervention study, using a random single blind controlled type trial, conducted at a pharmacy in Elche on female clients with mild alterations in their lipid profile. Since they were patients with a high cardiovascular risk, the investigators aimed to determine the effect of the administration of (FS+Y+D), (Y+D) and (D) on various nutritional indicators.

A monitoring of nutritional intervention was carried out for 30 days and blood samples were obtained by capillary puncture for total cholesterol levels, triglycerides, glucose. These parameters were determined in situ by dry chemistry. A series of anthropometric measures were also carried out at the beginning and at the end of the study including weight and height, BMI (Body Mass Index), WHR (waist-hip ratio), systolic and diastolic arterial pressure and heart rate.

Statistical analysis was carried out using STATGRAPHICS Centurion XV software (StatPoint Technologies, Inc. Warrington, VA, USA); likewise, significance was defined at p ≤ 0.05. Data are reported as mean ± standard error of the mean (sem). Intra-group statistical comparisons were performed using the following hypothesis tests, both parametric and non-parametric: t-test, sign test and signed rank test for paired samples. Inter-group statistical comparisons were performed using the one-way analysis of variance and the Kruskal-Wallis hypothesis tests. Also, Fisher's least significant difference (LSD) Multiple Range Test and Tukey's honestly significant difference (HSD) were used in order to determine which means were significantly different from the others. In addition, Generalized Multiple Regression was used to statistically analyze the relationships between the variations in the lipid profile and the different factors included in the study.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily participation
* ages between 25-70 years
* undergoing dislipidemia
* with no pharmacological treatment
* cholesterol (250-300 mg/dL)
* triglycerides (160-175 mg/dL)

Exclusion Criteria:

* subjects undergoing any pharmacological treatment that may influence lipid metabolism
* lipid levels outside the range of those specified in the inclusion criteria
* subjects that were deemed to be unlikely to complete the treatment or to cooperate fully at the investigator´s discretion.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Anthropometric characteristics of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  In this table we present five parameters of the three intervented groups

CONTACTS AND LOCATIONS:
Overall Officials: Elena García, PDI, Principal Investigator — Universidad Miguel Hernandez de Elche
Locations (1):
- Pharmacy Iborra Campos, Elche, Alicante, Spain